CLINICAL TRIAL: NCT04403958
Title: The Use of Proximal Carpal Row Versus Iliac Crest Bone Graft in Total Wrist Fusion - a Randomized Controlled Multicenter Trial Comparing Two Operative Techniques (PROOF II - Trial)
Brief Title: The Use of Proximal Carpal Row Versus Iliac Crest as Bone Graft in Total Wrist Fusion
Acronym: PROOF II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Töölö Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Kymenlaakso Central Hospital Kotka Finland (Other)
Responsible Party: Principal Investigator, Samuli Aspinen, Principal investigator, Töölö Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1467/2020
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Wrist Arthritis; Fusion; Joint
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRC (Experimental): Total wrist arthrodesis with PRC and dorsal plate
  Interventions: Procedure: PRC
- TWA (Active Comparator): Total wrist arthrodesis with dorsal plate
  Interventions: Procedure: TWA

INTERVENTIONS:
Procedure: PRC — Total wrist arthrodesis with dorsal plate using proximal row of the wrist as bone graft
  Arms: PRC
Procedure: TWA — Total wrist arthrodesis with dorsal plate using iliac crest as bone graft
  Arms: TWA

SUMMARY:
Study purpose is to compare the outcome after total wrist arthrodesis (TWA) with proximal carpal row (Proximal Row Carpectomy = PRC) as bone graft versus iliac crest cancellous bone graft.

Patients with radiologically and clinically confirmed advanced osteoarthritis are randomized (1:1 computer generated sequence with random block size) to two parallel groups and will undergo either total wrist arthrodesis with PRC or TWA with iliac crest bone grafting.

Baseline data is collected preoperatively and is a follow-up visits at every 6 weeks after the surgery is arranged until the wrist is fused. The primary end-point is 6 months and the primary outcome is fusion rate.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75
* Symptom duration > 3 months
* American Society of Anaesthesiologists physical status (ASA) I-III
* Fluent in written and spoken Finnish

Exclusion Criteria:

* Age <18 or >75 years
* Rheumatoid arthritis
* Heavy smoking (> 20 cigarettes per day)
* Condition or medication affecting bony healing (eg diabetes mellitus with poor glycemic control, malnutrition, use of per oral corticosteroids)
* Ulnar variance > 1 mm
* Wrist pain treatable with partial wrist fusion
* Previous partial wrist fusion
* Alcohol or drug abuse
* Neurological condition affecting upper limb function
* Less than 6 months after another operation of the same upper limb

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Fusion rate (percent) | 6 months

SECONDARY OUTCOMES:
Pain (Visual Analogue Scale) | 6 months
  The VAS is derived by health care professional question of pain in scale 0 to 100 mm (0 mm =no pain, 100 mm =worst possible pain)
Patient-Rated Wrist Evaluation (PRWE) | 6 months
  The PRWE comprises 15 questions to measure wrist pain and disability in daily activities. In PRWE patients rate wrist pain and disability from 0 to 10 and it consists two subscales: Pain and Function (0=best possible outcome, 10=worst possible outcome)
Quick-Disabilities of the Arm, Shoulder and Hand (QuickDASH) | 6 months
  The QuickDASH is self-reported questionnaire and shortened version of DASH outcome measure to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb in 11 dimensions in 1-5 scale (1=best possible outcome, 5=worst possible outcome)
Global improvement | 6 months
  Global rating to treatment effect will be evaluated by question: "How would you rate the function of your hand compared to the situation before the treatment?". The options are in 5-step Likert scale from (-2) Much worse to (+2) Much better
Grip strength | 6 months
  Grip strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in kg and percentage of the unaffected side
Operative time | Perioperative
  Operative time is measured in minutes for time in the operation theatre and time used for surgery
Complications | 12 months
  Incidence of complications (i.e. non-union, fracture, re-operation, infection, hematoma, iatrogenic tendon/nerve/arterial injury, complex regional pain syndrome) is recorded and compared between study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Samuli Aspinen, M.D., Ph.D., Principal Investigator — HUS Töölö Hospital

IPD SHARING:
Plan to Share IPD: No